CLINICAL TRIAL: NCT02430064
Title: Effects of Chronic Intake of Processed Foods on Circulating Inflammatory Markers in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Responsible Party: Principal Investigator, Clett Erridge, Research Fellow, University of Leicester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CE01
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low PAMP diet then high PAMP diet (Experimental): All subjects on study proceed from 7 days low PAMP diet to 4 days high PAMP diet
  Interventions: Other: Low PAMP diet

INTERVENTIONS:
Other: Low PAMP diet

SUMMARY:
This study aims to investigate the effects of diets enriched or depleted in foods at high risk of containing pro-inflammatory bacterial molecules, on markers of inflammation and cardiometabolic risk in healthy men. The study design is an interventional diet study, with 7 days dietary advice to avoid processed foods, followed by 4 days in which lunch and evening meal are provided to volunteers. Anthropometric and blood markers of cardiovascular disease risk are measured at the start and end of each dietary phase. The aim is to gain an improved understanding of how processed foods modify risk of cardiometabolic disease.

DETAILED DESCRIPTION:
This study aims to investigate the effects of diets enriched or depleted in foods at high risk of containing pro-inflammatory bacterial molecules, on markers of inflammation and cardiometabolic risk in healthy men. The study design is an interventional diet study, with 7 days dietary advice to avoid processed foods, followed by 4 days in which lunch and evening meal are provided to volunteers. Anthropometric and blood markers of cardiovascular disease risk are measured at the start and end of each dietary phase. The aim is to gain an improved understanding of how processed foods modify risk of cardiometabolic disease.

Three blood samples, each of 15 ml, will be taken on days 0, 8 and 12. Measurements at each timepoint include weight, waistline, serum low-density lipoprotein cholesterol, high density lipoprotein cholesterol, triglycerides, insulin, leptin, C-reactive protein and endotoxin.

Volunteers will be requested to avoid processed foods, ready-prepared meals, foods containing minced meats, foods containing ready-chopped vegetables, cheese or chocolate for the first 7 days of the study.

For days 8 to 11, volunteers will be provided with meals, purchased from local supermarkets, which from previous tested were found to contain high levels of bacterial pro-inflammatory molecules (PAMPs).

Diet diaries collected during the study will be combined with diet recall information to investigate habitual and on-study frequency of consumption of specific food groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male consenting volunteers
* Age 18-60

Exclusion Criteria:

* Any existing inflammatory condition, such as chronic kidney disease, inflammatory bowel disease, coronary artery disease or rheumatoid arthritis
* Evidence of an infection within the last two weeks
* Users of prescription medications
* Vaccination within the last two weeks

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Serum C-reactive protein and white blood cell counts will be used as markers of inflammation (composite). | up to 11 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Clett Erridge, PhD, Principal Investigator — University of Leicester

REFERENCES:
- [Derived] Herieka M, Faraj TA, Erridge C. Reduced dietary intake of pro-inflammatory Toll-like receptor stimulants favourably modifies markers of cardiometabolic risk in healthy men. Nutr Metab Cardiovasc Dis. 2016 Mar;26(3):194-200. doi: 10.1016/j.numecd.2015.12.001. Epub 2015 Dec 19. PMID 26803597